CLINICAL TRIAL: NCT05196230
Title: A Virtual Dental Office Experience for Children With Autism Spectrum Disorder - A Pilot Randomized Controlled Trial
Brief Title: A Virtual Dental Office Experience for Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Azadeh Kushki, Senior Scientist, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: eREB#209
Record Dates: First submitted 2021-06-25; First posted 2022-01-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Condition (360° Video) (Experimental): The 360° video (experimental) group will be mailed a study tablet with the 360° video prior to the dental visit.
  Interventions: Device: Experimental Condition (360° Video)
- Control Condition (Social Story) (Active Comparator): The treatment-as-usual (control) group will be mailed a study tablet with a social story prior to the dental visit.
  Interventions: Device: Control Condition (Social Story)

INTERVENTIONS:
Device: Control Condition (Social Story) — The control condition is a social story, which is treatment as usual for preparing clients for their initial visit at Holland Bloorview's dental clinic. The control condition will be delivered through the study tablet. The investigators will ask parents to read it to their child once a day for the week leading up to their appointment. If the child is reading on their own, the investigators will request that parents be in the room with participants while they are. The social story takes approximately five minutes to read.
  Other Names: Treatment as usual
  Arms: Control Condition (Social Story)
Device: Experimental Condition (360° Video) — The 360° video is from the point of view of a seated dental client and the participant will be able to explore the scene around them (navigating through the tablet's touch screen). The simulation will include scenes/features that may be anxiety-provoking for some participants. These will include loud noises commonly encountered in the dentist's office (e.g. tooth brushing, dental drills), as well as social stimuli (e.g. the dental clinician), and new environments (e.g., the dental visit room). The investigators will ensure that participants understand that they can stop at any time (e.g., if they are feeling anxious or overwhelmed), and the investigators will ask parents to explore the 360° video with their child for the week leading up to their appointment.
  Arms: Experimental Condition (360° Video)

SUMMARY:
The objective of this study is to evaluate the effectiveness of virtual reality (360° video) compared to a social story for reducing pre-visit dental anxiety for children with autism spectrum disorder (ASD) improve the dental visit experience for children, their families, and clinicians. The secondary objective is to perform a cost comparison analysis of the 360° video product as compared to a social story for Holland Bloorview's dental clinic.

DETAILED DESCRIPTION:
Participation in this research study will include daily at-home use of either the 360° video (experimental condition) or social story (control condition) for seven days prior to participant's first visit to the dental clinic, as well as parent, child, and dental clinician questionnaires. Both pre-visit experiences will be delivered remotely, in-home, and through the use of a study-provided tablet. Participants will be asked to access the pre-visit experience exclusively through use of the study-provided tablet, and to document daily use of the tablet experience on a Daily Journal log provided to families with the tablet. Tablets will have the assigned pre-visit experience pre-loaded (360° video or social story) and will be locked with a passcode, to ensure that participants do not engage with the tablet or pre-visit experience prior to 7-days before their dental visit. Tablets and pre-visit questionnaires will be mailed out to families two weeks prior to their onsite dental appointment. One week plus one business day prior to their initial dental visit at Holland Bloorview, families will be contacted by telephone to provide them with the tablet passcode so participants can access their assigned pre-visit experience (360° video or social story) and to remind them of the study protocol. Parents can be provided with a copy of the instructions by email as well if participants prefer, however, tablet passcodes will only be provided over the telephone.

Randomization This will be a single-blinded study, whereby participants will know which experimental group participants have been allocated to, but the dental clinician will not. Research study staff will also be aware of participant allocation.

Experimental Condition (360° Video) The 360° video has been developed by Shaftesbury Films in consultation with Holland Bloorview dental, research study staff, and family advisors. The 360° video is from the point of view of a seated dental client and the participant will be able to explore the scene around them (navigating through the tablet's touch screen). The simulation will include scenes/features that may be anxiety-provoking for some participants. These will include loud noises commonly encountered in the dentist's office (e.g. tooth brushing, dental drills), as well as social stimuli (e.g. the dental clinician), and new environments (e.g., the dental visit room). The investigators will ensure that participants understand that they can stop at any time (e.g., if participants are feeling anxious or overwhelmed), and the investigators will ask parents to explore the 360° video with their child.

Control Condition (Social Story) The control condition is a social story, which is treatment as usual for preparing clients for their initial visit at Holland Bloorview's dental clinic. As for the experimental condition, the control condition will be delivered through the study tablet. The investigators will ask parents to read it to their child once a day for the week leading up to their appointment. If the child is reading on their own, the investigators will request that parents be in the room with participants. The social story takes approximately five minutes to read.

PRE-DENTAL VISIT

Parent Questionnaires One week plus one business day prior to dental visit, parents will receive a reminder call (and email, if requested) from study staff. This will be to provide families with the tablet passcode and remind them to fill out the questionnaires and of the pre-visit experience protocol. Parents will be asked to fill out questionnaires characterizing their child prior to their onsite dental visit. The questionnaires will collect information on the following domains: demographic and prior dental experience (Demographic and Prior Experience Questionnaire), child's sensory profile (Short Sensory Profile (SSP)), anxiety (Screen for Anxiety Related Disordered (SCARED)), ASD symptomatology (Social Communication Questionnaire (SCQ)), and any co-morbidities (Child Behaviour Checklist (CBCL)). Questionaries will be mailed to participants two weeks prior to their dental visit, along with the study tablet. Parents will be asked to bring the complete questionnaires and study tablet with them to their dental visit to return to study staff. If parents fail to return study tablet and/or questionnaires, staff will provide them with prepaid and labelled shipping envelopes for the study tablet and/or questionnaires to be returned in the mail.

DAY OF DENTAL VISIT

Research families will be asked to come to Holland Bloorview 30-minutes ahead of their scheduled appointment time with the dental clinic. Research study staff will be waiting at Reception for the family to check in, at which point participants will provide the family with the questionnaire to fill out and invite participants to put on the smartwatch.

Smartwatch (Physiological Signal Recording) Participants will be asked to wear a Samsung Galaxy smartwatch to record time-stamped heart rate (electrocardiogram) and accelerometry signals. The functionality of the smartwatch will be restricted for study purposes (user cannot launch apps or change settings). The smartwatch will record continuously from the time it is put on the participant until it is taken off by study staff in the waiting room at the end of their visit. Study staff will indicate on the watch (set a 'marker') when the participant is beginning their dental visit (upon leaving waiting area). As an exploratory aim, the investigators will examine the change in physiological indices (average heart rate, heart rate variability) before and during the dental visit obtained from the smartwatch.

Participant Questionnaire Participants will be asked to fill out a brief questionnaire to assess their level of pre-visit anxiety (State-Trait Anxiety Inventory - for Children (STAI-CH) "How I Feel Questionnaire"). As the investigators are not excluding participants based on cognitive or verbal abilities, STAI-CH can be filled out with the help of a parent, if needed.

POST-DENTAL VISIT

Clinician Questionnaire The dental clinician will be required to fill out a post-visit questionnaire at the end of the participant's dental visit to assess visit completeness (progression through 5-steps). This questionnaire also contains one question assessing the participant's behavior (Frankl behavior rating scale), and two questions regarding blinding: the first probes whether or not the participant/family disclosed their group allocation; the second asks the clinician to guess which group they believed the participant was allocated to.

Parent Questionnaires Parents will be asked to complete a brief custom follow-up questionnaire after their child's dental appointment, assessing their provision of the pre-visit experience to their child over the past week and their experience traveling to Holland Bloorview for their dental appointment. This questionnaire will be conducted by study staff with parents within two business days of their dental appointment, by telephone or Zoom, as preferred. If the parent wishes to complete the follow-up questionnaire with study staff immediately following their child's dental appointment, they will be able to. Study staff will schedule the follow-up questionnaire with parents in the dental waiting area before their child's dental appointment.

ELIGIBILITY:
Inclusion Criteria:

* A community diagnosis of ASD
* Aged 4-12
* First time client of Holland Bloorview dental (has not previously received dental services at Holland Bloorview dental)
* Dental appointment at least 3 weeks away from time of initial contact
* Parent-predicted difficulty for child to sit through entire dental appointment

Exclusion Criteria:

• Parent predicts no difficulty for child to sitting through entire dental appointment

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Dental visit "completeness" | During the dental appointment
  The investigators will compare the difference in the number of children who complete each stage of the appointment between the two intervention groups using the clinician-rated, post-visit questionnaire. This questionnaire assesses a five-step checklist of visit completeness (1 = Waiting room, 2 = Sitting in dental chair, 3 = Teeth counting, 4 = Teeth cleaning, and 5 = Fluoride painting).

SECONDARY OUTCOMES:
Pre-visit anxiety | Immediately preceding dental appointment
  A state anxiety measure (State-Trait Anxiety Inventory for Children, Form C-1) will be used to assess between group differences in pre-visit anxiety. Higher scores indicate greater state anxiety (minimum score = 20, maximum score = 60).

OTHER OUTCOMES:
Heart rate | During dental appointment
  As an exploratory aim, the investigators will examine participant's physiological (heart rate) response during the dental visit to see if there is a difference in arousal between group allocations. The investigators will examine average heart rate and heart rate variability both before (in the waiting room) and during the participant's dental visit. Physiological arousal will be measured using a smartwatch (Samsung Galaxy Watch).
Cost comparison analysis | through study completion, an average of 1 year
  The investigators will carry out a cost comparison analysis of the 360° video compared to current practice (a social story). The main target of the cost comparison analysis is the cost per dental treatment for both the dental clinic and the client (participant). This will be established based on (1) number of visits required to complete a given treatment (in this instance, routine cleaning) and (2) cost per visit.

CONTACTS AND LOCATIONS:
Overall Officials: Azadeh Kushki, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada